CLINICAL TRIAL: NCT07120724
Title: Efficacy and Safety of Chinese Medicine in the Treatment of Chikungunya Fever: A Real-World Observational Study
Brief Title: Real-World Study on Chinese Medicine for Treating Chikungunya Fever
Status: Recruiting | Type: Observational
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ZE2025-299-01
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chinese Medicine Group: Intervention: Patients receive only TCM treatments, which may include herbal formulas (e.g., decoctions, granules) or acupuncture, tailored to their syndrome differentiation (e.g., heat-clearing, detoxifying, or dampness-resolving therapies).
- Western Medicine Group: Intervention: Patients receive only standard Western medical care, which may include antipyretics (e.g., acetaminophen), NSAIDs for pain, and supportive treatments (e.g., hydration).
- Integrated Therapy Group: Intervention: Patients receive both Chinese and Western treatments.

SUMMARY:
This study aims to evaluate the effectiveness and safety of Chinese Medicine-used alone or combined with Western medicine-in treating chikungunya fever, a mosquito-borne viral disease causing fever, rash, and severe joint pain. With recent outbreaks in China (including over 3,000 cases in Foshan, Guangdong) and no specific antiviral treatment available, Chinese medicine may offer a valuable therapeutic option based on its symptom-relief and syndrome-specific approach.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the suspected or confirmed diagnostic criteria for chikungunya fever;
2. Symptom onset ≤3 days before enrollment;
3. Actual prescribed treatment aligns with the study's group assignment (TCM, Western medicine, or combined therapy)
4. Signed informed consent form

Exclusion Criteria:

1. Severe chikungunya fever;
2. Participation in another drug clinical trial within the past 3 months;
3. Any other condition deemed by the investigator as unsuitable for enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants will be selected from patients affected by the chikungunya fever outbreak in Foshan, Guangdong Province, with current concentration in Shunde District.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Change in Rash Severity Assessed by Modified Eczema Area and Severity Index (mEASI) | From the enrollment to the end of the observation on the 28th day
  Quantifies absolute change from baseline in skin inflammation severity using a modified Eczema Area and Severity Index (mEASI) scoring system.(Higher scores indicate more severe inflammation)
Proportion of Participants Achieving Clinically Significant Improvement in Joint Symptoms Assessed by Disease Activity Score 44 (DAS44) | From enrollment to the end of the observation on the 28th day.
  Measured by the Disease Activity Score 44 (DAS44) scale, which evaluates:
  * 44 swollen joint counts
  * 44 tender joint counts
  * Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)
  * Patient's global health assessment (VAS 0-100 mm)
  Scoring range: 0-10
  * Lower scores indicate better disease control
  * Clinically significant improvement defined as:
    * 1.2 point reduction from baseline AND Final DAS44 score ≤3.2
Time to Complete Fever Resolution | From the enrollment to the end of the observation on the 28th day.
  Records the duration (in hours/days) from treatment initiation until the patient achieves sustained normal body temperature (≤37.3°C) without antipyretics.

SECONDARY OUTCOMES:
Time to Viral RNA Clearance (RT-PCR Negative) | From the enrollment to the end of the treatment on the 5th day.
  Measures the days required for chikungunya virus RNA to become undetectable in blood by RT-PCR.
Proportion of participants with normalized blood cell counts | From the enrollment to the end of the treatment on the 5th day.
  Percentage of subjects achieving restoration of white blood cell, lymphocyte and platelet counts to normal reference ranges
Time to Symptom Recovery | From the enrollment to the end of the observation on the 28th day.
  Assesses the duration until complete resolution of all symptoms (e.g., fatigue, headache, myalgia).
Incidence of Complications | From the enrollment to the end of the observation on the 28th day.
  Monitors the occurrence of complications (e.g., chronic arthritis, neurological involvement, secondary infections).
Adverse Events (AEs) | From the enrollment to the end of observation on the 28th day.
  Records all AEs (e.g., allergic reactions, gastrointestinal issues) and their relation to the treatment.
Proportion of participants with normalized C-reactive protein (CRP) levels | From the enrollment to the end of the treatment on the 5th day.
  Percentage of subjects achieving serum CRP levels within normal reference range (≤5 mg/L)
Proportion of participants with restored baseline-abnormal coagulation parameters | From the enrollment to the end of the treatment on the 5th day.
  Percentage of subjects achieving normalization in coagulation parameters that were abnormal at baseline (e.g., PT, aPTT, INR, D-Dimer)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form: Study Protocol (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT07120724/Prot_ICF_000.pdf